CLINICAL TRIAL: NCT01071941
Title: rRp450-Phase I Trial in Liver Metastases and Primary Liver Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: Kenneth K. Tanabe, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Kenneth K. Tanabe, MD, Chief, Surgical Oncology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-042; 5R21CA119600 (NIH)
Record Dates: First submitted 2010-01-13; First posted 2010-02-19 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Liver Metastases; Primary Liver Cancers
Keywords: rRp450; Herpes virus; Gene therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental): The first subjects will receive a single infusion of rRp450. Subsequent subjects will receive rRp450 as four doses administered every 1-2 weeks.
  Interventions: Biological: administration of rRp450 into the hepatic artery

INTERVENTIONS:
Biological: administration of rRp450 into the hepatic artery — Administration of rRp450 into the hepatic artery either as a single infusion, or as four infusions administered every one to two weeks.
  Other Names: rRp450

SUMMARY:
The purpose of this research study is to determine the safety of rRp450 and the highest dose of this agent that can be given to people safely. We are also looking to see how well the body tolerates the study agent, how the agent is absorbed by the liver cancers, how quickly the agent is eliminated from the body, and what kind of anti-cancer effect it may have. rRp450 is a type of gene therapy and a form of the Herpes simplex virus 1 (or HSV). HSV is a virus that usually causes cold sores of the mouth. In extremely rare circumstances, this virus can cause severe infections, such as an infection of the brain. rRp450 was developed from an HSV and specially altered to target and kill cancer cells.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of the study agent that can be administered safely without severe or unmanageable side effects in participants that have liver tumors, not everyone who participates in this research study will receive the same dose of the study drug. The dose the participant receives will depend on the number of participants who have been enrolled in the study before and how well they tolerated their doses.
* Depending upon when the participant enrolls in this study, they will either receive a single injection of rRp450, or up to 4 weekly injections of rRp450. Participants in both groups will be monitored after the rRp450 injection in the hospital and in the clinic. As of July, 2013, because the first phase of the study has been completed, all participants from here forward will receive 4 weekly injections of rRp450
* For the rRp450 injection, we will insert a small tube into the artery that supplies blood to the liver. rRp450 will be injected into this tube so it goes directly to the liver. Another tube is inserted into the blood vessel that drains blood from the liver. We will use this tube to take blood samples to monitor how the body absorbs and breaks down rRp450.
* After the rRp450 injection, participants will be monitored closely for any side effects. Vital signs will be closely monitored before, during and after rRp450 injection. After the rRp450 injection, the tubes are removed.
* The following tests and procedures are done before the rRp450 injection: determination of overall health condition, performance status evaluation, review of current medications and any side effects, physical exam and vital signs.
* The following tests and procedures will be done during the injection of rRp450: vital signs, review of any side effects, research blood samples taken from a vein in your arm, and research blood samples taken from your liver vein.
* The following tests and procedures will be done after rRp450 injection: 1 Hour after; blood tests: 6 and 12 hours after; blood tests, vital signs, routine blood tests, samples of saliva and swabs of the skin of the penis or vaginal secretions (hour 12 only): 24 hours after, Between days 4 to 7 and Between days 10 to 14; review of current medications and side effects, physical exam, vital signs, routine blood tests, swab samples of saliva, blood test to see if the body has produced antibodies against HSV-1 (only on day 4 to 7 and only for participants enrolled in the single injection group).
* Liver and tumor biopsies will be performed about 6 days after the rRp450 injection.
* Participants will be asked to return to the clinic 2 weeks, 4 weeks, and every 3 months thereafter after their last injection of study medication.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more and able to understand and sign a written informed consent form
* Histologically confirmed diagnosis of cancer with liver metastases, or histologically confirmed primary liver cancer (e.g. hepatocellular carcinoma, cholangiocarcinoma, or gallbladder carcinoma). Subjects may have extrahepatic spread of malignancy, except they may not have brain metastases. Subjects with a history of more than one invasive malignancy remain eligible for this study, but in these instances, a liver biopsy is required to document the histology of the liver tumor. An exception to this criterion is made for basal cell carcinoma.
* Subjects must have primary or metastatic liver malignancies which are surgically unresectable, and exhausted all standard therapeutic options
* Patients with hepatocellular carcinoma must have received sorafenib as one of the standard treatment options prior to being enrolled into the study
* No liver surgery (including radiofrequency ablation), chemotherapy (including bevacizumab), immunotherapy, or liver radiotherapy within 4 weeks of enrollment.
* ECOG performance status 0, 1 or 2 and life expectancy of greater than 12 weeks based on the investigator's clinical judgment.
* Serum hematology and chemistry test results as outlined in the protocol.
* Tumor volume occupies less than 50% of liver by volume as assessed by CT scan or MRI scan within 4 weeks of treatment
* Negative pregnancy test (serum or urine) in premenopausal women
* Prior exposure to HSV-1 as determined by blood test

Exclusion Criteria:

* Clinical or pathological diagnosis of cirrhosis, hemachromatosis, or heptic fibrosis
* Ascites or complete occlusion of main portal vein
* Hepatitis C infection, chronic infection with hepatitis B, infection with HIV, or evidence of hepatic insufficiency
* Inability to practice contraception with condoms as prescribed by the protocol
* Active infection requiring treatment with systemic antibiotics or systemic anti-fungal agents
* Being treated with immunosuppressive agents such as systemic corticosteroids or cyclosporine
* Unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia, or need for antiarrythmic medication for which inability to take an oral preparation of regular medication for 48 hours would represent an unacceptable risk.
* Known existing uncontrolled coagulopathy, hemorrhagic disorder, or inability to discontinue coumadin or plavix for 5 days prior to each treatment (except for prophylaxis against portacath-associated thrombosis, which does not require cessation of therapy).
* History of seizures
* Allergy to acyclovir or inability to receive contract for CT and MRI scans
* Prior liver resection of greater than 2 anatomic segments as defined by Couinaud (subjects that have undergone prior liver wedge excisions or segmental resections are not excluded on this basis alone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of rRp450 administered into the hepatic artery as a single dose. | 3 years
Evaluate the safety and tolerability of rRp450 administered into the hepatic artery as four doses administered every 1-2 weeks. | 3 years
Determine the dose-limiting toxicities and maximum dose of rRp450 that can be safely administered into the hepatic artery when administered weekly for four doses. | 3 years
Characterize rRp450 pharmacokinetics and viral shedding. | 3 years

SECONDARY OUTCOMES:
Assess the relationship between systemic rRp450 levels and clinical toxicity. | 3 years
Evaluate tumor biopsies for rRp450 replication, tumor response and immune cell infiltrates. | 3 years
Correlate radiographic and pathologic assessments of tumor response. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K. Tanabe, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States